CLINICAL TRIAL: NCT03661450
Title: Evaluation of the Accuracy of a Clinical Decision-Support System (CDSS) to Support Detection of SIRS and Sepsis in Paediatric Intensive Care Patients Compared to Medical Specialists
Brief Title: Evaluation of CDSS in Detection of SIRS and Sepsis in Pediatric Patients
Acronym: CADDIE2
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: Technische Universitaet Braunschweig (Other); Helmholtz Centre for Infection Research (Other)
Responsible Party: Sponsor
Other Study IDs: 7804_BO_S_2018
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: SIRS; Sepsis; Pediatric SIRS
Keywords: Clinical Decision-Support System
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PICU-Patients: Pediatric patients admitted after 01.08.2018
  Interventions: Diagnostic Test: Clinical Decision-Support System

INTERVENTIONS:
Diagnostic Test: Clinical Decision-Support System — Patient Data is evaluated by a Clinical Decision-Support System searching for age-adapted pediatric SIRS-criteria, aiming for a high sensitivity and specificity

SUMMARY:
This trial aims to evaluate the accuracy of a Clinical Decision-Support System to support early recognition of SIRS in paediatric intensive care patients. This assessment will be rated by the primary goals, the sensitivity and specificity of the system. Two experienced paediatric intensivists, who are blinded for the CDSS results, will analyse the electronic patient file (EPF) for SIRS criteria and thus establish our Goldstandard. All SIRS events recognized by the CDSS during the patient's stay are taken into account and will be compared with the established Goldstandard.

The secondary goal of this trial is to evaluate the CDSS-results with the assessment of SIRS by paediatric doctors during their routine work on the PICU.

DETAILED DESCRIPTION:
Clinical decision-support systems (CDSS) are designed to solve knowledge-intensive tasks for supporting decision-making processes. Although many approaches for designing CDSS have been proposed, due to high implementation costs, as well as the lack of interoperability features, current solutions are not wellestablished across different institutions. Recently, the use of standardized formalisms for knowledge representation as terminologies as well as the integration of semantically enriched clinical information models, as openEHR Archetypes, and their reuse within CDSS are theoretically considered as key factors for reusable CDSS. The investigators already successfully transferred their concept into a prototype and evaluated the practicability on clinical data sets and in close cooperation between the clinicians and the technical experts. To the author's knowledge, currently, there are no openEHR based CDSS approaches which have been implemented and evaluated with such complex and important clinical contexts. Hence, the first clinically evaluated CDSS based on openEHR was successfully designed. When enhancing the described approach and implementing a live system, it might support clinicians to identify the patient's course of disease at an early stage, which can lead to better outcome for the patient. Furthermore, the system can serve as a basis for integrating (cross-institutional) machine learning components that could facilitate dealing with other high-complex decision problems or revealing yet unknown disease patterns.

ELIGIBILITY:
Inclusion Criteria:

* all pediatric patients admitted to our PICU

Exclusion Criteria:

* patients that are supposed to stay for less than 12 hours on our PICU

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients from newborn to young adults up to 18 years that are admitted to our PICU, there is a wide range from infectious causes, post-operative-care of pediatric surgery, cardiac surgery, organ-transplants etc, newborns connatal syndromes and organdysplasia.
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of CDSS compared to Goldstandard | 8 months
  Assessment of sensitivity and specificity of a CDSS compared to Goldstandard established by two independed blinded paediatric intensivists, the analysis will be done with Wald-Confidence interval and comparison of the lower limit of the confidence interval with the defined range of the null hypothesis.

SECONDARY OUTCOMES:
Sensitivity and specificity of CDSS on daily level | 8 months
  Evaluation of sensitivity and specificity of the CDSS on daily levels compared with the Goldstandard with respect to correlation of days within one patient's course with general estimating equations.
Comparison of CDSS with assessment of MDs taking care of the patients | 10 months
  Evaluation of sensitivity and specificity of the CDSS on daily level and patient level compared with recognition of SIRS by paediatric doctors during daily routine with McNemar testing and general estimating equations.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marschollek, PhD, Study Chair — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Wulff A, Montag S, Rubsamen N, Dziuba F, Marschollek M, Beerbaum P, Karch A, Jack T. Clinical evaluation of an interoperable clinical decision-support system for the detection of systemic inflammatory response syndrome in critically ill children. BMC Med Inform Decis Mak. 2021 Feb 18;21(1):62. doi: 10.1186/s12911-021-01428-7. PMID 33602206
- [Derived] Wulff A, Montag S, Steiner B, Marschollek M, Beerbaum P, Karch A, Jack T. CADDIE2-evaluation of a clinical decision-support system for early detection of systemic inflammatory response syndrome in paediatric intensive care: study protocol for a diagnostic study. BMJ Open. 2019 Jun 19;9(6):e028953. doi: 10.1136/bmjopen-2019-028953. PMID 31221891